CLINICAL TRIAL: NCT01167660
Title: Non Invasive Measurement of Coagulation in Term and Preterm Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pag-ThM2
Record Dates: First submitted 2010-07-05; First posted 2010-07-22 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2010-06

CONDITIONS: Blood Coagulation Tests
Keywords: Coagulation tests; Neonates; Non invasive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy newborn babies: Healthy newborn babies immediately after birth.
  Interventions: Device: The Thrombo-Monitor (ThM)
- Sick newborn babies: Sick newborn babies whose medical condition indicates performing coagulation tests.
  Interventions: Device: The Thrombo-Monitor (ThM)

INTERVENTIONS:
Device: The Thrombo-Monitor (ThM) — Non-invasive measurement of coagulation status and comparison to standard blood coagulation tests. In healthy neonates - immediately after birth, before the administration of vitamin K. Coagulation tests will be done on an umbilical cord blood sample. In sick neonates, coagulation studies will be done according to the medical condition.

SUMMARY:
The purpose of this study is to assess the reliability of a new non-invasive device to assess the blood coagulation status among term and preterm babies.

DETAILED DESCRIPTION:
Coagulation abnormalities among neonates aren't common - but can be life threatening. Testing the coagulation system in small babies involves drawing significant amounts of blood (especially in premature babies). Non-invasive testing can help assess and treat term and preterm neonates at risk. Recently, a non-invasive device to assess the blood coagulation status was developed - The Thrombo-Monitor (ThM). The objective of this study is to assess the reliability of this new non-invasive device among term and preterm babies by comparing the result of the ThM reading to coagulation analysis from blood.

ELIGIBILITY:
Inclusion Criteria:

* Newborn babies - term and preterm
* Written parental informed consent

Exclusion Criteria:

* Congenital anomalies / chromosomal abnormalities

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term and preterm babies born in Meir Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Reliability of the non-invasive ThM device. | From birth up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ita Litmanovitz, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel